CLINICAL TRIAL: NCT06877910
Title: Deciphering the Molecular Traits of Non-canonical Responders to Advance Personalized Therapy in Gastric Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1377/20(2378)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective, identification set: A workflow based on numerous statistical analyses will assign the individual molecular outcomes in one of the three categories considered (exceptional responders, conventional responders, fast progressors). The information retrieved with this first level of analysis will be summarized in a single tool for the prediction of individual risk (nomogram). In order to guarantee reproducibility, the prognostic classifier will be obtained from a retrospective cohort of patients with mGC treated with standard first-line chemotherapy.
- Prospective, validation set: Definition of the evolutionary trajectories of atypical responders mGC, by taking blood samples from patients enrolled in the prospective cohort, collected at predefined time points. The serial collection of blood samples will allow the study of circulating nucleic acids (cfTNA, liquid biopsy) for the monitoring of genomic alterations and for the levels of gene expression differentially represented in exceptional responders and fast progressors.

SUMMARY:
Retrospective-prospective observational study in which a novel whole-exome sequencing (WES) approach will be used in association with whole-transcriptome sequencing (WTS) to analyze two independent and equally sized cohorts of patients with mGC.

DETAILED DESCRIPTION:
A workflow specifically designed for this project will be adopted, using clinical outcomes as a benchmark for comparative analyses, to generate a molecular classifier applicable to all patients affected by metastatic gastric cancer mGC and predict atypical tumor responses. Molecular features differently represented in exceptional responders and fast progressors will be monitored by liquid biopsy in patients included in cohort B, consisting of a validation set, leveraging a high-sensitivity technological level that allows to detect both genomic alterations and expression at the transcription level.

In addition, CSCs isolated from fast progressors will be studied with over 1,000 antitumor agents to discover vulnerabilities not currently known.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Histological diagnosis of locally advanced or metastatic gastric cancer (GC) or gastroesophageal junction carcinoma (EJC);
* Adequate biological material for molecular analysis, collected (at surgery or by biopsy) before the administration of any anti-tumor treatment (chemotherapy and/or radiotherapy);
* ECOG PS 0-2;
* Adequate hematological, hepatic and renal function;
* Measurable disease according to RECIST criteria;
* Written informed consent.

Exclusion Criteria:

* Previous chemotherapy for metastatic disease;
* Comorbidities not controlled with adequate medical therapy;
* Brain metastases;
* Patient unable to give adequate consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic inoperable GC who are candidates for first-line chemotherapy and who meet the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival PFS | 5 years
  PFS will be defined as the time from the start of first-line chemotherapy to disease progression or death

SECONDARY OUTCOMES:
Overall survival OS | 5 years
  OS will be defined as the time from the start of first-line chemotherapy to death (from any cause)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer institute, Rome, Italy